CLINICAL TRIAL: NCT05122234
Title: Effectiveness and Safety Profile of Mesenchymal Stem Cell Secretomes as a Treatment for Severe Cases of COVID-19
Brief Title: Mesenchymal Stem Cell Secretome In Severe Cases of COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Murdani abdullah, Prof. M.D., PhD, FACG, FASGE, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 54/FI/P-KCOVID-19.2B3/IX/2020
Record Dates: First submitted 2021-11-13; First posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
Keywords: Severe Covid-19; secretome; mesenchymal stem cell; cytokine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Secretome - mesenchymal stem cell group (n = 20) (Experimental): This group will be given secretome - mesenchymal stem cell and COVID-19 standard therapy
  Interventions: Biological: Injection of secretome - mesenchymal stem cell; Drug: Standard treatment of Covid-19
- Control ( n= 20) (Placebo Comparator): This group will be given placebo and COVID-19 standard therapy
  Interventions: Other: Placebo; Drug: Standard treatment of Covid-19

INTERVENTIONS:
Biological: Injection of secretome - mesenchymal stem cell — Secretome will be given once at a dose of 15 ml per administration dissolved in 100 ml of normal saline. The administration is done intravenously for 60 minutes.
  Arms: Secretome - mesenchymal stem cell group (n = 20)
Other: Placebo — Normal saline
  Arms: Control ( n= 20)
Drug: Standard treatment of Covid-19 — Standard treatment of Covid-19 based on national protocol.

SUMMARY:
This study is a multi-centre randomized controlled trial involving severe covid-19 patients. The intervention group will receive mesenchymal stem cell secretomes and standard covid-19 therapy, while the control group receive placebo and standard covid-19 therapy. Clinical presentation, inflamatory marker, laboratory and radiological parameters, RT-PCR conversion, safety profile, and mortality rate will be monitored for a maximum of 14 days after intervention.

ELIGIBILITY:
Inclusion Criteria:

1. All individuals aged 18 to 65 years
2. It has been confirmed positive for COVID-19 by throat swab / sputum / brochoalveolar lavage (BAL) with real-time reverse transcription polymerase chain reaction (RT-PCR)
3. Categorized as a severe case of COVID-19 patient
4. Agree to participate and sign the informed consent

Exclusion Criteria:

1. History of allergy to penicillin, streptomycin, and amphotericin-B
2. Have any cancer conditions
3. Active in other intervention studies
4. Have had other intervention studies in the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-11-14 (Actual)

PRIMARY OUTCOMES:
Assessment of inflamation marker levels | Day 0 (before intervention), day 7, day 14
  The inflamatory marker assessed in this study is IL-6, IL-10, LIF, VEGF, and Ferritin. The inflamatory marker level will assess on day 0 (before intervention), day 7 after intervention, and day 14 after intervention.

SECONDARY OUTCOMES:
Assessment of clinical outcome | before and after intervention (maximum 14 days after intervention)
  Clinical outcome assessed in this study were body temperature, oxygen saturation, respiratory rate, shortness of breath, cough, and phlegm on cough.
Assessment of laboratory routine | before and after intervention (maximum 14 days after intervention)
  Laboratory routine assessed in this study is NLR, lymphocyte count, thrombocytes count, CRP, blood gas analysis, bilirubin, albumin, SGOT, SGPT, ureum/creatinin, glomerular filtration rate (GFR), electrolyte, myoglobin, troponin, D-dimer.
Assessment of photo thorax | before and after intervention (maximum 14 days after intervention)
  Photo thorax will assess before and after intervention
Assessment of RT-PCR conversion | before and after intervention (maximum 14 days after intervention)
  RT-PCR conversion will assess before and after intervention
Mortality rate | maximum 14 days after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Murdani Abdullah, Prof. M.D., PhD, FACG, FASGE, Principal Investigator — Departemen of Internal Medicine, Faculty of Medicine, University of Indonesia
Locations (4):
- Indonesia (4):
  - RSUP Fatmawati, Jakarta, DKI Jakarta
  - RSUP Persahabatan, Jakarta, DKI Jakarta
  - RSUPN Dr. Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta
  - Rumah Sakit Universitas Indonesia, Depok, West Java